CLINICAL TRIAL: NCT03293511
Title: Oxytocin Modulates Eye Gaze Behavior During Social Processing and Associations With Trait Autism
Brief Title: Oxytocin Modulates Eye Gaze Behavior During Social Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESCT_neuSCAN_42
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Oxytocin; Eye tracking; Autistic trait

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind within-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order of administration: oxytocin - placebo (Experimental): Participants first receive oxytocin (24 IU). After a washout period of 2 weeks, they receive placebo nasal spray
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo
- Order of administration: placebo - oxytocin (Experimental): Participants first received placebo nasal spray. After a washout period of 2 weeks, they then receive oxytocin (24 IU).
  Interventions: Drug: intranasal oxytocin; Drug: intranasal placebo

INTERVENTIONS:
Drug: intranasal oxytocin — 24 IU of oxytocin nasal spray will be applied to each subject.
Drug: intranasal placebo — 24 IU of of placebo nasal spray will be applied to each subject.

SUMMARY:
The main aim of the study is to examine whether the effects of intranasal oxytocin on eye-gaze behavior towards social stimuli are modulated via individual differences in trait autism

DETAILED DESCRIPTION:
In this double-blind, within subject, placebo controlled design a total of n = 40 healthy male subjects will receive either 24 IU of oxytocin or placebo (interval between administration > two weeks). 45 minutes after treatment subjects will undergo a total of 7 eye-tracking paradigms examining eye-gaze behavior during social processing: (1) dynamic social-nonsocial visual preference task during which movies of dynamic geometric images (DGI) and dynamic social images (DSI) will be presented; (2) non-biological versus biological motion task; (3) social attention and motivation of sharing enjoyment; (4) preference for emotional faces versus schematic faces (emoticons); (5) shared social attention - shared gaze direction with an actor shifting his attention to different objects; (6) preferred visual scanning of face regions in emotional faces; and, (7) eye gaze in response to empathy eliciting visual stimuli. Autistic and associated traits will be assessed using the Autism Spectrum Quotient (ASQ), Social Responsibilities Scale (SRS) and the Interpersonal Reactivity Index (IRI). Within-subject differences in the effects of oxytocin on social eye gazing behaviour will be related to individual differences in autistic traits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury
* Visual impairments
* Use of medication
* Contraindications for oxytocin administration

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Global eye gaze characteristic: differences between oxytocin and placebo treatment | 45-90 minutes after treatment administration
  Global eye-gaze patterns will be compared between the administration of oxytocin and placebo
Feature-specific eye gaze characteristics: differences between oxytocin and placebo treatment | 45-90 minutes after treatment administration
  Localized feature-specific eye gaze patterns will be compared between oxytocin and placebo treatment

SECONDARY OUTCOMES:
Global eye gaze characteristic - associations with autism traits | 45-90 minutes after treatment administration
  Within-subject differences in global eye gaze characteristics between the oxytocin and placebo administration will be examined for associations with individual differences in autism traits
Feature-specific eye gaze characteristics - associations with trait autism | 45-90 minutes after treatment administration
  Within-subject differences in localized feature-specific eye gaze characteristics between the oxytocin and placebo administration will be examined for associations with individual differences in autism traits

CONTACTS AND LOCATIONS:
Overall Officials: Juan Kou, MSc, Study Chair — University of Electronic Science and Technology of China
Locations (2):
- China (2):
  - school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan
  - University of Electronic Science and Technology of China, Chengdu, Sichuan

REFERENCES:
- [Derived] Le J, Kou J, Zhao W, Fu M, Zhang Y, Becker B, Kendrick KM. Oxytocin Facilitation of Emotional Empathy Is Associated With Increased Eye Gaze Toward the Faces of Individuals in Emotional Contexts. Front Neurosci. 2020 Aug 11;14:803. doi: 10.3389/fnins.2020.00803. eCollection 2020. PMID 32848571